CLINICAL TRIAL: NCT01063985
Title: A Comparison of Skin Prick Tests, Clinical Symptoms and Nasal Challenge Using a New Mouse Extract
Brief Title: A Comparison of Skin Prick Tests, Clinical Symptoms, and Nasal Challenge Using a New Mouse Extract
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Allison Norton, MD and Ryszard Dworski, MD, Vanderbilt University Medical Center
Other Study IDs: 091213
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Mouse Allergies; Mouse Sensitization
Keywords: Skin testing for mouse allergies

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to test a new mouse skin test extract on people who work with mice in a lab or through animal care. It has a higher level of the major allergen and therefore may be better at diagnosing mouse allergies in this population.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to mouse on a regular basis through occupation or animal care. Patients must sign informed consent before completing any study procedure.
* Healthy subjects age >18 years and <60 years
* Females with no child bearing potential. Females are considered not to have child bearing potential before their menarche, at least 2 years after menopause or if they have had a total hysterectomy or bilateral oophorectomy
* Females with child bearing potential if they fulfill the following criteria: Use of a medically accepted contraceptive method (hormone birth control [orally, injectable, or implant for at least 2 months prior to enrollment], intrauterine device, spermicide used with a male condom, bilateral tubal ligation, diaphragm with spermicide, female condom), and have a negative pregnancy test
* Patients who are able to understand the information given, be compliant with the protocol including investigational product administration and visit schedules as well as recording information requested by the investigators.

Exclusion Criteria

* Present history of tobacco smoking (within the past 12 months or ex-smoker with >10 pack years).
* Illicit drug use.
* Asthma requiring treatment with medications other than beta-2 inhaled agonists and leukotriene inhibitors.
* Patients with a history of asthma or wheezing with an FEV1 <80%
* Subjects who have taken a nasal adrenergic agonist the day of the procedure
* Use of H1 antagonists, leukotriene inhibitors, tricyclic antidepressants, phenothiazines, nasal antihistamines, or ocular antihistamines within 5 days prior to the testing.
* Subjects who are on nasal, oral steroids, or ketotifen within 2 weeks of the procedure
* Subjects taking beta blockers, ace inhibitors, continuous systemic corticotherapy, immunosuppressive drugs, reserpine, clonidine or monoamine oxidase inhibitors.
* Patients who have received any desensitization for mouse allergen in the past 5 years
* Ongoing immunotherapy with any other allergen.
* Patients with any nasal condition that could confound the efficacy or safety assessments, for example nasal polyposis, nasal ulcers, nasal surgery 6 weeks prior to study or tumors.
* Patients with any past or current clinically significant condition that may affect the patient's participation or the outcome of the study to the discretion of the investigator. These include, but are not limited to, anaphylaxis with cardio-respiratory symptoms (to any known or unknown source including mice exposure), chronic urticaria and angioedema unless related to mouse exposure, severe atopic dermatitis, malignancy, cardiovascular, hepatic, renal, hematological, neurological, immunological, and endocrine disease.
* Hyper responsiveness to glycerin control on nasal challenge as defined by a non-cumulative score of 5 on the nasal challenge symptom score.
* Although fetal risk is not expected to be high, women of childbearing potential who may be pregnant or who are not on adequate contraceptives will be excluded from the study (as defined in inclusions). In addition pregnant or breastfeeding women will also be excluded from the study.
* Study staff, investigators, sub-investigators, as well as their children or spouses and family members of all study staff should not be enrolled in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals between the ages of 18-60 who are exposed to mice through occupation or animal care.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine the optimal concentration of mouse extract based on the skin prick test using the nasal challenge and clinical symptoms to confirm their true mouse allergic status in a sample of people exposed to mice. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Ryszard Dworski, MD, Principal Investigator — Vanderbilt University; Allison Norton, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Clinical Research Center at Vanderbilt University, Nashville, Tennessee, United States